CLINICAL TRIAL: NCT05196074
Title: Airway Closure During Extracorporeal Membrane Oxygenation: The AiCLOSE Study
Acronym: AiCLOSE
Status: Recruiting | Type: Observational
Sponsor: Lorenzo delSorbo (Other)
Collaborators: Unity Health Toronto (Other)
Responsible Party: Sponsor-Investigator, Lorenzo delSorbo, MD, Critical Care Medicine Department, Toronto General Hospital, University Health Network, Toronto
Organization: University Health Network, Toronto (Other)
Other Study IDs: 21-5784
Record Dates: First submitted 2021-12-15; First posted 2022-01-19 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Acute Hypoxemic Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute hypoxemic respiratory failure patients on VV-ECMO
  Interventions: Other: Acute hypoxemic respiratory failure patients on VV-ECMO

INTERVENTIONS:
Other: Acute hypoxemic respiratory failure patients on VV-ECMO — To describe the prevalence of complete airway closure in patients with acute hypoxemic respiratory failure on VV-ECMO and its association with outcome.

SUMMARY:
About 65,000 Canadians develop acute respiratory failure requiring breathing machines (ventilators) to give oxygen to their lungs. Unfortunately, up to 50% of these individuals will not survive their illness.

Mechanical ventilation through breathing machines, though potentially lifesaving, may further injure the lungs and the respiratory muscles. In the patients with the most severe and life threatening forms of respiratory failure a breathing machine alone may not be able to provide enough oxygen to the lungs and vital organs. In these critical situations, patients may require an artificial lung machine, which is referred to as extracorporeal membrane oxygenation (ECMO) to temporarily replace the function of the patient's own lung and supply critical oxygen to the body, while protecting the damaged lungs. How to use the breathing machine safely while a patient is on ECMO is still unknown. Using conventional breathing machine settings while on ECMO can lead to large portions of the lungs or airway to remain collapsed, which can contribute to further lung damage.

The investigators have recently discovered a way of detecting if patients on a breathing machine suffer from collapsed airways. Knowing if the most severe patients on ECMO have airway collapse is a pivotal question that the investigators plan to answer in our study. The investigators will use our technique to determine how many patients on ECMO have airway closure and determine if this contributes to a longer time on ECMO and a longer time on a breathing machine, and if this impacts a patient's survival in the intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Acute hypoxemic respiratory failure
* VV-ECMO
* Less than 24 hours from ECMO cannulation

Exclusion Criteria:

* Air leak
* VV-ECMO as bridge to lung transplantation
* Status asthmaticus

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Acute hypoxemic respiratory failure patients on VV-ECMO.
Sampling Method: Non-Probability Sample
Enrollment: 299 (Estimated)
Dates: Start 2022-04-04 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Prevalence of complete airway closure | Day 1 of VV-ECMO cannulation
  Prevalence of complete airway closure during day 1 of VV-ECMO support.

SECONDARY OUTCOMES:
Correlation of airway closure with patient outcomes | Up to 90 days from VV-ECMO cannulation
  Evaluation of the correlation between the presence of complete airway closure and the level of airway opening pressure and both clinical and physiological outcomes listed below:
  a. Clinical outcomes i. duration of ECMO support at 90 days ii. duration of mechanical ventilation at 90 days iii. ICU mortality iv. mortality at 90 days v. prevalence of barotrauma vi. daily ECMO support I. sweep gas II. Flow vii. Daily fluid balance b. Physiological outcomes i. time to recovery I. In spontaneous modes of ventilation compliance will be measured by dividing tidal volume by driving pressure ii. time to protective spontaneous breathing (defined as: a. ventilator not continuously triggered by the patient I. Pocc is measured by performing an end-expiratory occlusion maneuver, freezing the ventilator waveform and measuring the drop in airway pressure.
  iii. lung recruitability iv. right ventricular dysfunction
Correlation of the degree of mismatch between clinical PEEP and AOP with patient outcomes | Up to 90 days from VV-ECMO cannulation
  Evaluation of the correlation between the degree of mismatch between clinical PEEP and AOP and patient outcomes listed below:
  a. Clinical outcomes i. duration of ECMO support at 90 days ii. duration of mechanical ventilation at 90 days iii. ICU mortality iv. mortality at 90 days v. prevalence of barotrauma vi. daily ECMO support I. sweep gas II. Flow vii. Daily fluid balance b. Physiological outcomes i. time to recovery I. In spontaneous modes of ventilation compliance will be measured by dividing tidal volume by driving pressure ii. time to protective spontaneous breathing (defined as: a. ventilator not continuously triggered by the patient I. Pocc is measured by performing an end-expiratory occlusion maneuver, freezing the ventilator waveform and measuring the drop in airway pressure.
  iii. lung recruitability iv. right ventricular dysfunction
Assessment of the distribution of airway closure within the lung and between the two lungs | Up to 90 days from VV-ECMO cannulation
  Assessment of the distribution of airway closure within the lung and between the two lungs by EIT.
Assessment of predictors of airway closure | Up to 90 days from VV-ECMO cannulation
  Assessment of body mass index and the degree of obesity as predictors of airway closure.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Del Sorbo, MD, Principal Investigator — University Health Network, Toronto; Laurent Brochard, MD, Principal Investigator — Unity Health Toronto; Michael Sklar, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No